CLINICAL TRIAL: NCT02459691
Title: Culturally-adapted Diabetes Prevention Lifestyle Intervention for Latinos in Primary Care (E-LITE Latinos)
Brief Title: Culturally-adapted Diabetes Prevention Lifestyle Intervention for Latinos (E-LITE Latinos)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Palo Alto Medical Foundation (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency); University of Illinois at Chicago (Other); University of Pittsburgh (Other); RTI International (Other); University of California Santa Cruz (Other)
Responsible Party: Principal Investigator, Jun Ma, MD, PhD, Beth and George Vitoux Professor of Medicine, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 14-10-365
Record Dates: First submitted 2015-05-29; First posted 2015-06-02 (Estimated); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: Prediabetic State; Metabolic Syndrome X; Insulin Resistance
Keywords: prediabetes; metabolic syndrome; lifestyle; behavior change; primary care; latinos; diet; physical activity
MeSH Terms: conditions — Prediabetic State; Metabolic Syndrome; Insulin Resistance; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Usual Care Only (Active Comparator): Patients assigned to this group will continue medical care as usual.
  Interventions: Other: Usual Care Only
- Vida Sana (Experimental): Patients assigned to this group will continue medical care as usual and in addition will receive the culturally adapted intervention.
  Interventions: Behavioral: Vida Sana

INTERVENTIONS:
Behavioral: Vida Sana — Vida Sana is a Diabetes Prevention Program-based, culturally-adapted intervention that will have 2 distinct stages: The intensive treatment stage will implement a culturally adapted year-long Group Lifestyle Balance curriculum. The curriculum uses a goal-based approach to promote positive outcome expectancies and foster self-efficacy. The maintenance stage will be focused on (1) facilitating continued behavior change; (2) fostering participants' self-efficacy and independence; and (3) reinforcing problem-solving and behavior maintenance skills. These will be done via secure e-messaging.
  Arms: Vida Sana
Other: Usual Care Only — Patients assigned to this group will continue medical care as usual. That is, they will continue to see their primary care provider and any specialist he/she may recommend. They may also access additional health education resources available at the Palo Alto Medical Foundation. They will continue to receive general age and gender-appropriate reminders of health maintenance tests/exams and immunizations, per Palo Alto Medical Foundation standard practice.
  Arms: Usual Care Only

SUMMARY:
The purpose of the study is to develop a culturally adapted intervention (CAI) program to improve weight and physical activity in overweight or obese adult Latinos at high risk for developing type 2 diabetes and/or cardiovascular disease (CVD) and to rigorously evaluate the effectiveness and implementation potential of the CAI program.

DETAILED DESCRIPTION:
This study has two phases: Phase 1: Formative research and Phase 2: Randomized Controlled Trial (RCT). The purpose of the formative research phase is to develop a culturally adapted intervention (CAI) program to improve weight and physical activity in overweight or obese adult Latinos at high risk for developing type 2 diabetes and/or cardiovascular disease (CVD). The purpose of the RCT is to rigorously evaluate the effectiveness and implementation potential of the CAI program.

The proposed intervention will uniquely adapt the coach-led, technology-supported Group Lifestyle Balance (GLB) program that the investigators proved effective in the investigators' prior trial called E-LITE, to provide culturally and linguistically appropriate lifestyle intervention for weight loss and increased physical activity among high-risk Latinos in primary care. The CAI will be delivered in small groups as well as using existing, rapidly expanding internet and mobile technologies (Website, email, and mobile text messaging). Once developed the investigators will subject the CAI to rigorous evaluation in an RCT of 186 eligible and consenting Latinos. The investigators hypothesize that CAI participants will achieve a greater mean reduction in body mass index (BMI) from baseline to 24 months (primary outcome) than usual care controls. Secondary outcomes will include measures of cardiometabolic risk factors (e.g., lower fasting glucose and lipid levels), psychosocial well-being (e.g., improved mood), and behavior change (e.g., increased physical activity). The overarching research goal is to determine the effectiveness and implementation potential of the CAI based on the Reach, Effectiveness, Adoption, Implementation, and Maintenance (RE-AIM) framework.

ELIGIBILITY:
Inclusion criteria:

* Age(as of date of enrollment):

  * Lower age limit: 18 years
  * Upper age limit: NONE (only exclude for cause, e.g. disease and functional limitations, as detailed below)
* Race/ethnicity: Mexican Latino of any race
* Gender: men and women
* Body mass index: ≥24 kg/m2 (≥22 kg/m2 if of Asian descent)
* Having pre-diabetes, metabolic syndrome, or both based on the following criteria:
* Pre-diabetes according to any one of the following criteria:
* Fasting plasma glucose of 100 to 125 mg/dL or HbA1c of 5.7 to 6.4 if detected by a recent (within the past year), documented, blood-based diagnostic test or by a fasting blood test during study screening
* Plasma glucose measured 2 hours after a 75 gm glucose load of 140 to 199 mg/dl if detected by a recent (within the past year), documented, blood-based diagnostic test (Oral glucose tolerance test will not be performed for study screening considering participant burden)
* Clinically diagnosed gestational diabetes mellitus during a previous pregnancy (may be self-reported)
* Metabolic syndrome according to 3 or more of the following:

  * Waist circumference ≥40 inches in men and ≥35 inches in women (≥35 inches in men and ≥31 inches in women, if of Asian descent)
  * Triglycerides >150 mg/dL
  * High-density lipoprotein cholesterol (HDL-C) <40 mg/dL in men and <50 mg/dL in women
  * Systolic blood pressure ≥130 mmHg or diastolic blood pressure ≥85 mmHg
  * Fasting plasma glucose of 100 to 125 mg/dL
* Primary Care Physician approval of patient contact for study screening
* Able and willing to enroll and provide informed consent, i.e., to meet the time and data collection requirements of the study, be randomized to one of two study arms, participate in follow-up for 24 months, and authorize extraction of relevant information from the Electronic Health Record.

Exclusion criteria:

* Medical exclusions:
* Previous diagnosis of diabetes (other than during pregnancy) or diabetes diagnosed as a result of fasting blood glucose or hemoglobin A1c levels obtained through study screening;
* Diagnosis of cancer (other than non-melanoma skin cancer) that is/was active or treated with radiation or chemotherapy within the past 2 years;
* Serious medical condition anticipated to prevent person from walking 1 mile (e.g., severe pulmonary disease or aortic stenosis)
* Severe medical co-morbidities that require aggressive treatment: e.g., stage 4 or greater renal disease, class III or greater heart failure, unstable coronary artery disease, liver or renal failure;
* Diagnosis of a terminal illness and/or in hospice care;
* Diagnosis of bipolar disorder or psychotic disorder within the last 2 years, or currently taking a mood stabilizer or antipsychotic medication
* Initiation or change in type or dosing of antidepressant medications within 2 months prior to enrollment (The patient will be re-contacted for a later cohort once his/her regimen has been stable for at least 2 months unless the person declines to participate altogether.)
* Have had or plan to undergo bariatric surgery during the study period
* Other exclusions:
* Inability to speak, read or understand Spanish or English
* Having no reliable telephone service
* Having no regular Internet access via a computer and/or mobile device (e.g., smart-phone)
* Currently pregnant or lactating or planning to become pregnant during the study period
* Plan to move out of the area during the study period
* Family/household member of another study participant or of a study staff member
* Investigator discretion for clinical safety or protocol adherence reasons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 191 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2019-05 (Actual); Study Completion 2019-05 (Actual)

PRIMARY OUTCOMES:
Change in weight from baseline | 12- and 24-months
  Change in weight

SECONDARY OUTCOMES:
Change in composite measure of cardiometabolic risk factors | Baseline, 12- and 24-months
  Blood pressure, waist circumference, waist-to-height ratio
Change in Body Mass Index from Baseline | 12- and 24-months
  BMI
Clinically significant weight loss | 12 and 24 months
  5% or greater weight loss

CONTACTS AND LOCATIONS:
Overall Officials: Jun Ma, MD, PhD, Principal Investigator — UIC

REFERENCES:
- [Derived] Rosas LG, Lv N, Xiao L, Lewis MA, Venditti EMJ, Zavella P, Azar K, Ma J. Effect of a Culturally Adapted Behavioral Intervention for Latino Adults on Weight Loss Over 2 Years: A Randomized Clinical Trial. JAMA Netw Open. 2020 Dec 1;3(12):e2027744. doi: 10.1001/jamanetworkopen.2020.27744. PMID 33337491
- [Derived] Rosas LG, Lv N, Xiao L, Lewis MA, Zavella P, Kramer MK, Luna V, Ma J. Evaluation of a culturally-adapted lifestyle intervention to treat elevated cardiometabolic risk of Latino adults in primary care (Vida Sana): A randomized controlled trial. Contemp Clin Trials. 2016 May;48:30-40. doi: 10.1016/j.cct.2016.03.003. Epub 2016 Mar 16. PMID 26995280